CLINICAL TRIAL: NCT01069523
Title: Electrophysiological Effects of Guanfacine Extended-Release (GXR) on Inhibitory Control in Children With Attention Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Electrophysiological Effects of Guanfacine Extended Release in Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC2009-499H
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Disorder with Hyperactivity; Guanfacine; Event Related Potentials
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients will be started on 1 mg of guanfacine extended release matching placebo tablets at week 1. A physician blind to drug status will titrate the study medication in week 2-3 to a maximum of 4 mg (4 tablets).
  Interventions: Drug: Placebo
- Guanfacine Extended Release (Experimental): Patients will be started on 1 mg of guanfacine extended release at week 1. A physician blind to drug status will titrate the study medication in week 2-3 to a maximum of 4 mg (4 tablets).
  Interventions: Drug: Guanfacine Extended Release

INTERVENTIONS:
Drug: Guanfacine Extended Release — Guanfacine is an alpha-2A agonist which is given one a day. the dose range is 1-4 mg. It is a tablet.
  Other Names: Intuniv
  Arms: Guanfacine Extended Release
Drug: Placebo — Table that match the 1 mg Guanfacine Extended Release Tablet. They are dosed once a day.
  Arms: Placebo

SUMMARY:
All subjects with the study will be children (age 6-12) with Attention Deficit Hyperactivity Disorder (ADHD). After baseline assessment confirms the presence of ADHD, children will have an Event related potential (ERP) (a type of electroencephalogram [EEG]) study. After the baseline EEG, children will be randomized to either placebo or GXR for a 4-week, parallel groups trial. During this trial, dosing will be flexibly adjusted according to patient response or presence of side effects. The dosage will range from 1-4 mg. At the end of the four week trial, a follow up ERP study will be obtained.

DETAILED DESCRIPTION:
All subjects with the study will be children (age 6-12) with Attention Deficit Hyperactivity Disorder (ADHD). After baseline assessment confirms the presence of ADHD, children will have an Event related potential (ERP) (a type of electroencephalogram [EEG]) study. After the baseline EEG, children will be randomized to either placebo or GXR for a 4-week, parallel groups trial. During this trial, dosing will be flexibly adjusted according to patient response or presence of side effects. The dosage will range from 1-4 mg. At the end of the four week trial, a follow up ERP study will be obtained. Our hypotheses are: A) GXR will be superior to placebo at reducing symptoms of ADHD as measured by standardized clinical diagnostic tools by week 3 of treatment. B) Compared to placebo and pretreatment measures, GXR at week 4 of treatment will increase the amplitude of the right frontal N200 and frontal-central P300, and such changes will correlate with clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 years
* Meet criteria for Attention Deficit Hyperactivity Disorder

Exclusion Criteria:

* Do not meet criteria for Major Depression, Bipolar, Autism
* Talking any psychotropic medication for a condition other than ADHD
* History of epilepsy, severe head injury or loss of consciousness
* History of Intolerance to guanfacine

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Pliszka, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Dept. Of Psychiatry, University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4/2010 through 6/2011 primarily through flyers in child psychiatry clinics and by informing families who called the clinic intake line.
Pre-assignment Details: After diagnostic assessment and confirmation that subjects meet study criteria, subjects were scheduled for a baseline EEG and they performed the Stop Signal Task while ERP data was obtained. 42 subjects completed baseline evaluation,13 did not complete baseline EEG, leaving 29 to be randomized to drug
Period: Overall Study
Arm/Group | Placebo | Guanfacine Extended Release
Started | 13 | 16
Completed | 9 | 9
Not Completed | 4 | 7
Not completed — Withdrawal by Subject | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Guanfacine Extended Release | Total
Number analyzed (Participants) | 13 | 16 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 16 | 29
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 8.78 (1.8) | 7.8 (1.2) | 8.29 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 6 | 10 | 16
Region of Enrollment [Number; unit: participants]
  United States | 13 | 16 | 29

OUTCOME MEASURES:

1. Primary Outcome: Dupaul ADHD Rating Scale
Description: 54 point scales assessing ADHD symptoms in a dimensional manner. 0 is no ADHD symptoms while 54 is severe. A score of 18 or below is the normative range.
Time Frame: Baseline and Follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Guanfacine: Patients will be started on 1 mg of guanfacine extended release at week 1. A physician blind to drug status will titrate the study medication in week 2-3 to a maximum of 4 mg (4 tablets).
Arm/Group | Placebo | Guanfacine
Number analyzed (Participants) | 9 | 9
units on a scale | 31.4 (16.5) | 13.6 (9.7)

2. Secondary Outcome: Clinical Global Impression- Improvement
Description: Blinded clinician overall assessment of the child global improvement in behavior-1 is very much improved, 2-much improved, 3- minimally improved, 4 no change, 5-minimally worse, 6- much worse, 7- very much worse
Time Frame: Week 4 of study
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Pill placebo
- Guanfacine: Blinded guanfacine capsule
Arm/Group | Placebo | Guanfacine
Number analyzed (Participants) | 9 | 9
units on a scale | 3.0 (1.1) | 2.0 (0.5)

ADVERSE EVENTS:
Time Frame: Adverse events assessed at each visit covering the week prior
Description: Adverse events were spontaneously reported by patients
Arm/Group | Placebo | Guanfacine Extended Release
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/16
Other Adverse Events (participants affected / at risk) | 5/13 | 10/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | Guanfacine Extended Release (N=16)
Stomachache (Gastrointestinal disorders) | 1 (1) | 1 (1) — Self report by child or parent
Dizziness (General disorders) | 1 (1) | 1 (1) — Self report by parent or child
Sedation (General disorders) | 3 (3) | 5 (5) — Self report by parent or child
Fatigue (General disorders) | 0 (0) | 3 (3) — Self report by parent or child

LIMITATIONS AND CAVEATS:
The intent of the study was to examine ERP waveforms associated with impulse control. Unfortuanately, the Stop signal task and EEG proved very difficult for this young group of subjects. The ERP data could not be fully analyzed and is not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No